CLINICAL TRIAL: NCT06371430
Title: A Randomized, Double-Blind Clinical Human Trial , Bone Bioactive Liquid Efficiency in Improving Implant Osteointegration and Oral Soft Tissue Helling
Brief Title: Bone Bioactive Liquid Efficiency in Improving Dental Implant Osteointegration Oral Soft Tissue Hellingand Oral Surgery
Acronym: BBLIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biointelligent Technology Systems SL (Industry)
Collaborators: Universidad Pública de Navarra (Other); Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Maher Atari Abouasi, Director, Biointelligent Technology Systems SL
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Biointelligent Technology Syst
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Wound Healing Disorder; Wounds and Injuries; Wound Surgical
Keywords: Bone bioactive liquid; Dental implant; Oral wound healing
MeSH Terms: conditions — Wounds and Injuries; Surgical Wound | interventions — Tooth Extraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain Scale (Placebo Comparator): To assess the efficacy of the surgical procedure, pain scale evaluations were conducted on day 1,4 and 7, following the surgery. This evaluation involved a direct contact with the patients to gauge their subjective pain experience. A modified visual analog scale (VAS) was utilized, as described in reference [34]. No pain scale = 0, moderate pain scale = 5 and maximum pain scale = 10 [21]. In addition to efficacy measurements, safety measurements were also considered. The occurrence of adverse events (AEs) and serious adverse events (SAEs) was monitored throughout the duration of the study. These events were either detected by the investigator or reported by the patients themselves. The aim was to identify any potential complications or issues that arose because of the surgical procedure.
  Interventions: Device: Dental Implant insertion and tooth extraction
- RFA and ISQ measurements (Placebo Comparator): After the implants were fully seated, a Smartpeg specific to the implant system and restorative platform diameter was used for each implant. RFA was then performed using an OsstellMentor device from Ostell/Integration Diagnostics in Gothenburg, Sweden. This analysis was used to measure the ISQ values for all implant surfaces at days 0, 7 and 30 post-surgeries. For each implant, 4 readings were taken per lingual, mesial, distal, and vestibular direction. The average ISQ values of all the readings were recorded. Following the RFA measurements, new sterile healing abutments were inserted, and the incisions were sutured to close the wounds.
  Interventions: Device: Dental Implant insertion and tooth extraction
- CBCT analysis (Experimental): CBCTs were captured for implants from six patients with total of 24 implants, with 12 implants Galaxy TS (non-treated) on one side of the jaw and 12 implants Galaxy TSA (treated with BBL) on the other side of the jaw. All patients in this group had implants inserted in the upper jaw and each patient had 4 implants inserted (All on 4 technique). The CBCTs scans were conducted at days 1 and 60 post-surgeries using a 3D Accuitomo 170 scanner (J. MORITA EUROPE GMBH). The scans were performed with the following technical parameters: 90 kV, 5 mA, 87.5 mAs, voxel size ranging from 125-250 µm, 360° rotation, and scanning time of 17.5 s as previously described [32]. To ensure accuracy, a bite mark was utilized during CBCT scanning to correspond to the patients' midline. Consistency in bite mark placement was maintained to ensure that the same slice was obtained for each scan performed on the patient
  Interventions: Device: Dental Implant insertion and tooth extraction

INTERVENTIONS:
Device: Dental Implant insertion and tooth extraction — The osteotomies were carried out at a speed of 800 rpm, using sequential burs of similar diameter for both the maxilar and the mandibular side. The drilling protocols followed the recommendations provided by the manufacturer, the Galaxy-Ziacom implant system, for standard drilling.
  The insertion of the implants was initiated using a motor handpiece at a speed of 20-50 rpm, without irrigation. The installation process was completed using a manual surgical torque wrench indicator. The maximum torque value (Ncm) reached at the end of implant insertion was recorded as the insertion torque (IT). A total of 264 implants were inserted in 33 patients, 160 implants were post-extraction and 104 implants were inserted after at least one-month post-extraction. The sutures were typically removed 1 week after the surgery, during the postoperative follow-up appointment.

SUMMARY:
The investigators implanted 264 Galaxy TS implants (with or without BBL) in 33 patients across both jaws. Implant stability and osseointegration were assessed using Initial Stability Quotient (ISQ) measurements, computed tomography (CBCT) scans and pain evaluations at various intervals post-surgery. Further, implant surfaces were examined using scanning electron microscopy (SEM) and atomic force microscopy (AFM). In vitro studies evaluated the efficacy of BBL on dental pulp pluripotent stem cells (DPPSCs) osteogenesis, and inflammatory factor modulation in human macrophages.

DETAILED DESCRIPTION:
Ensuring implant stability and longevity is pivotal for patient satisfaction and quality of life. Our recent discovery, BBL, novel bone bioactive liquid, demonstrated promising properties in improving implant surfaces, alleviating pain, and expediting oral healing. In this multi-center randomized, double-blind clinical trial, investigators sought to evaluate the impact of BBL on the clinical performance of Galaxy TS implants.

Methods Investigators implanted 264 Galaxy TS implants (with or without BBL) in 33 patients across both jaws. Implant stability and osseointegration were assessed using Initial Stability Quotient (ISQ) measurements, computed tomography (CBCT) scans and pain evaluations at various intervals post-surgery. Further, implant surfaces were examined using scanning electron microscopy (SEM) and atomic force microscopy (AFM). In vitro studies evaluated the efficacy of BBL on dental pulp pluripotent stem cells (DPPSCs) osteogenesis, and inflammatory factor modulation in human macrophages.

ELIGIBILITY:
inclusion criteria:

* Age 18 years or older.
* sufficient residual bone volume to accommodate implant placement without requiring bone augmentation, minimum ridge height and width of ≥ 9mm and ≥ 6mm, respectively, and healed bone sites with a minimum of 1 months of post-extraction healing.

exclusion criteria

* Patients with alcoholism.
* Smoking habits.
* History of illicit drug use were excluded.
* Patients with heart diseases.
* Diabetes.
* Previous bone regenerative or augmentation procedures.
* Bleeding disorders.
* Compromised immune systems.
* History of radiation therapy
* Treatment with steroids or bisphosphonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
ISQ measurements | 3 month
  Implant stapelity

SECONDARY OUTCOMES:
CBCTs analysis | 2 month
  Quantify new bon formation

CONTACTS AND LOCATIONS:
Locations (1):
- Biointelligent Technology Syst, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided